CLINICAL TRIAL: NCT02466295
Title: The Comparison of the Effect of Pressure-controlled Ventilation and Volume-controlled Ventilation on the Gastric Insufflations in I-gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 4-2015-0280; NCT02425618 (obsolete NCT alias)
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: General Anesthesia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Volume-controlled ventilation (Experimental): The patient's lungs will be mechanically ventilated using the volume-controlled ventilation with tidal volume 8 ml/kg.
  Interventions: Other: Volume-controlled ventilation
- Pressure-controlled ventilation (Experimental): The patient's lungs will be mechanically ventilated using the pressure-controlled ventilation with tidal volume 8 ml/kg.
  Interventions: Other: Pressure-controlled ventilation

INTERVENTIONS:
Other: Volume-controlled ventilation — I-gel will be inserted into the patient's mouth. After confirmation of adequate ventilation with the i-gel, the patient's lungs will be mechanically ventilated using the volume-controlled mode with tidal volume 8 ml/kg during surgery.
  Arms: Volume-controlled ventilation
Other: Pressure-controlled ventilation — I-gel will be inserted into the patient's mouth. After confirmation of adequate ventilation with the i-gel, the patient's lungs will be mechanically ventilated using the pressure-controlled mode with tidal volume 8 ml/kg during surgery.
  Arms: Pressure-controlled ventilation

SUMMARY:
The purpose of this study is to investigate whether the pressure controlled ventilation can reduce gastric insufflation compared to the volume controlled ventilation in patients who were mechanically ventilated with the i-gel.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged over 20 yrs who are scheduled for surgery under general anesthesia

Exclusion Criteria:

* upper gastrointestinal surgery,
* surgery of long duration more than 4 hours,
* anticipated difficult intubation,
* body mass index more than 35 kg/m2,
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
gastric antral area | Within 5 minutes after the end of surgery
  The gastric antral area will be measured using ultrasonography.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, Seoul, South Korea